CLINICAL TRIAL: NCT06152965
Title: Functional Activity and Safety of a Food for Special Medical Purposes in Subjects Undergoing Bariatric Surgery: a Multicenter Prospective Observational Clinical Trial
Brief Title: Multivitamin Support Following Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Bioitalia srl (Industry)
Responsible Party: Sponsor
Other Study IDs: GS/01/19
Record Dates: First submitted 2023-11-17; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Bariatric Surgery
Keywords: VSG; RYGB; micronutrients deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Bariatric surgery (BS), an effective treatment for severe obesity and its comorbidities, may result in micronutrient and vitamin deficiencies. This monocentric prospective observational study aimed at evaluating the efficacy of a specifically designed vitamin/mineral formula (Bariatrifast) for preventing and treating micronutrient deficiencies in patients submitted to BS.

DETAILED DESCRIPTION:
Although BS effectively reduces body weight, improves metabolic alterations, and enhances overall health, it may also lead to micronutrients deficiency. This prospective observational study aimed at evaluating the effectiveness and safety of a specific FSMP (Food For Special Medical Purposes) in maintaining an adequate vitamin and micronutrient intake in patients with obesity submitted to VSG (Vertical Sleeve Gastrectomy) or RYGB (Roux-en-Y gastric bypass) . The included 20 consecutive patients with severe obesity who underwent BS (11 males, 9 females, all aged ≥18 years, with a BMI ≥ 40 kg/m2 or ≥ 35 kg/m2 with at least one obesity-related comorbidity, followed for one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* age >18yrs
* Written Informed consent done
* Bariatric surgery done

Exclusion Criteria:

* alcool or drugs abuse
* psychiatric illness
* allergy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational, prospective study included 20 consecutive patients with severe obesity who underwent BS (11 males, 9 females, all aged ≥18 years, with a BMI ≥ 40 kg/m2 or ≥ 35 kg/m2 with at least one obesity-related comorbidity. In the, 10 patients had hypertension, 5 insulin resistance, 5 type 2 diabetes, 2 non-alcoholic liver disease, 7 gastroesophageal reflux disease, 7 dyslipidemia and 2 obstructive sleep apnea. Ten of them underwent VSG and the other 10 RYGB. Patients were recruited at the Obesity and Lipodystrophy Center, University Hospital of Pisa
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy of Bariatrifast on vitamins concentration | One year. The study protocol included a presurgical visit (V0), and 4 follow up visits at 1 (V1), 3 (V2), 6 (V3), and 12 (V4) months after BS
  *25-OH Vitamin D3 in microgram/Liter (mcg/L) and vitamin B12 in nanogram/Liter (ng/L)

SECONDARY OUTCOMES:
evaluation of other parameters from blood test | One year. The study protocol included a presurgical visit (V0), and 4 follow up visits at 1 (V1), 3 (V2), 6 (V3), and 12 (V4) months after BS
  * Blood counts: red blood cells in number per microliter (10^6/microliter); hemoglobin in gram/liter (g/L); white blood cells in number per microliter (10^3/microliter); platelets in number per microliter (10^3/microliter)
  * ferritin in microgram/Liter (mcg/L),
  * ionized calcium in millimoles per liter (mmol/L),
  * PTH parathormone in nanogram/Liter (ng/L),
  * folic acid microgram/Liter (mcg/L), recorded at each visit
evaluation of body composition | One year. The study protocol included a presurgical visit (V0), and 4 follow up visits at 1 (V1), 3 (V2), 6 (V3), and 12 (V4) months after BS
  * Body weight (kilograms)

CONTACTS AND LOCATIONS:
Overall Officials: Ferruccio Santini, MD, Principal Investigator — Obesity and Lipodystrophy Center, University Hospital of Pisa (Italy)
Locations (1):
- Obesity and Lipodystrophy Center, University Hospital of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Basolo A, Bechi Genzano S, Vitti J, Salvetti G, Gilio D, Ceccarini G, Scartabelli G, Lippi C, Bellini R, Mancini R, D'Imporzano S, Moretto C, Angeli V, Troiani D, Fierabracci P, Jaccheri R, Calderone A, Poma AM, Chiovato L, Saponati G, Santini F. Efficacy of multivitamin support following bariatric surgery in patients with obesity: a prospective observational study. Eat Weight Disord. 2024 May 7;29(1):34. doi: 10.1007/s40519-024-01655-7. PMID 38714632